CLINICAL TRIAL: NCT02687386
Title: A Phase 1 Study of Intravenous EGFR-ErbituxEDVsMIT (EEDVsMit) in Children With Recurrent / Refractory Solid or CNS Tumours Expressing Epidermal Growth Factor Receptor (EGFR) (ECREST Study)
Brief Title: A Study of Intravenous EEDVsMit in Children With Recurrent / Refractory Solid or CNS Tumours Expressing EGFR
Acronym: ECREST
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study medication no longer in production
Sponsor: Dr David Ziegler (Other)
Collaborators: Engeneic Pty Limited (Industry)
Responsible Party: Sponsor-Investigator, Dr David Ziegler, Chief Investigator, Sydney Children's Hospitals Network
Organization: Sydney Children's Hospitals Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCA001
Record Dates: First submitted 2016-01-28; First posted 2016-02-22 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumours; CNS Tumours
Keywords: Recurrent; Refractory
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mitoxantrone packaged EDV (Experimental): Mitoxantrone packaged EDV (EnGeneIC Dream Vector)
  Interventions: Drug: Mitoxantrone packaged EDV (EnGeneIC Delivery Vehicle)

INTERVENTIONS:
Drug: Mitoxantrone packaged EDV (EnGeneIC Delivery Vehicle) — EnGeneIC Delivery Vehicles (EDVs) are nanocells which can be loaded with anti-cancer drugs (mitoxantrone in this study) and targeted to tumor cells. These bacterially-derived nanocells are coated in bispecific antibodies (BsAb) that recognize oncogenic receptors on the tumor cell surface. Once bound to the tumour cell, the targeted and drug-loaded EDVs are endocytosed and release their toxic payload to destroy the tumor cell.
  Other Names: EDV also stands for EnGeneIC Dream Vector

SUMMARY:
This is an open-label, sequential dose exploration study of single agent EEDVSMit administered by intravenous (IV) infusion twice weekly, followed by weekly maintenance dosing, in children with recurrent/refractory solid or CNS tumours.

DETAILED DESCRIPTION:
Eligible subjects enrolled in the study will receive EEDVSMit by IV injection twice weekly as a 20 min infusion beginning at study day 1 for the first cycle (4 weeks) then weekly for subsequent cycles. Subjects will undergo radiological assessment of their tumours after the first cycle, and every second cycle thereafter. Dosing with EEDVSmit will continue unless there is radiographic evidence of progressive disease (PD) per RECIST criteria version 1.1, the subject becomes intolerant to the study medication, signs and symptoms of clinical progression are evident as determined by the principal investigator, or the subject/parent/guardian withdraws consent. Suspected tumour progression should be confirmed with a repeat scan after 4 weeks to exclude the possibility of pseudoprogression.

Determination of EGFR expression for eligibility of subjects will be assessed at the local site. In addition, radiological assessment confirming measurable disease by the RECIST criteria is also required for entry into the Part B of the study.

The study will be conducted in two parts: Part A -Dose Exploration and Part B -Dose Expansion.

Part A - Dose Exploration:

The dose exploration part of the study is aimed at determining a recommended phase 2 dose (RP2D) in this patient group. A standard dose escalation with a rolling 6 design will be used.

Part A will commence dosing at one log scale below the maximum dose tested in the recent adult recurrent glioma trial (with the first 4 doses administered at 1/10 of the starting dose) and escalate to a maximum of 8x109 EEDVSMit evaluating the safety and tolerability, of EEDVSMit. The first 4 doses administered will be reduced by a further log reduction.

Part B - Dose expansion:

The dose expansion phase (Part B) will begin upon completion of the dose exploration (Part A). Up to 12 subjects with recurrent/refractory solid or CNS tumours will be treated at the Recommended Phase Two Dose (RPTD). All doses, including the first 4, will be at the same dose level established in Part A (RPTD).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 2 years and ≤ 21 years old at the time of study enrolment.
* Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age
* Patients must have relapsed or refractory solid or CNS tumours or have a diagnosis of DIPG. Patients must have had histologic verification of malignancy at original diagnosis or relapse, or a diagnosis of DIPG by MRI imaging.
* Patients must have either measurable or evaluable disease for Part B of the study only
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study.
* Any active uncontrolled infection
* Patients who are known to be serologically positive for Hepatitis A, B or C, or have a history of liver disease, other forms of hepatitis or cirrhosis.
* Known positive test for human immunodeficiency virus infection
* Patients with disease of any major organ system that would compromise their ability to withstand therapy
* Concurrent or prior (within 7 days of enrolment) anticoagulation therapy, except low molecular weight heparins or low dose aspirin
* Patients receiving corticosteroids must be on a stable dose that has not been increased for at least 7 days prior to study enrolment.
* Patients who are currently receiving another investigational drug are ineligible.
* Patients who are currently receiving other antineoplastic agents are ineligible.
* All herbal supplements, vitamins, and nutritional supplements taken within the last 30 days prior to dosing on Day 1 (and continued use, if appropriate), must be reviewed and approved by the Study Chair.
* Patient will not be available for protocol-required study visits or procedures, to the best of the subject/parent/guardian's and investigator's knowledge.
* Patient has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject/parent/guardian to give written informed consent and/or to comply with all required study procedures.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Patients will be screened for antibodies to S. typhimurium and will not be eligible until antibodies are non-detectable
* Patients will be screened for IL6 and TNFa cytokines and will not be eligible until levels are less than 3x times the detectable limit of the assay.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
MTD at which fewer than one third of patients experience dose limiting toxicity as assessed by CTCAE v4.0 | Day 28 (cycle 1)
  To determine a recommended phase 2 dose (RP2D) for EEDVsMit administered intravenously in children with recurrent / refractory solid or CNS tumours expressing EGFR
Incidence of treatment-related adverse events as assessed by CTCAE v4.0 | Up to 35 days after the completion of study treatment
  To define and describe the toxicities of EEDVSMit administered on these schedules in children with recurrent/refractory solid or CNS tumours
Incidence of all adverse events as assessed by CTCAE v4.0, clinically significant changes in vital signs, ECGs and clinical laboratory tests | Up to 35 days after the completion of study treatment
  Assess the safety and tolerability of EEDVSMit in children with recurrent/refractory solid or CNS tumours.

SECONDARY OUTCOMES:
Assess disease response according to RECIST version 1.1 for children with recurrent/refractory solid or CNS tumours | Up to 35 days after the completion of study treatment
  To preliminarily define the anti-tumour activity of EEDVSMit and assess response rates using RECIST version 1.1 criteria in children with recurrent/refractory solid or CNS tumours within the confines of a phase 1 study.
Assess overall survival | 12 months from the date the last subject was enrolled in the study.
  Assess overall survival (OS) in children with recurrent/refractory solid or CNS tumours treated with EEDVSMit on this schedule
Time to response assessed by radiological imaging and RECIST v1.1 | Evaluated at Day 56 (after cycle 2), then every second cycle to the end of study treatment (up to 12 months)
  Estimate the time to response.

CONTACTS AND LOCATIONS:
Overall Officials: David Ziegler, MBBS, Study Chair — Sydney Children's Hospitals Network
Locations (2):
- Australia (2):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data is planned to be shared with EnGeneIC.

REFERENCES:
- [Derived] Evans L, Walker R, MacDiarmid J, Brahmbhatt H, Anazodo A, McCowage G, Gifford AJ, Kavallaris M, Trahair T, Ziegler DS. A Phase 1 Study of Intravenous EGFR-ErbituxEDVsMIT in Children with Solid or CNS Tumours Expressing Epidermal Growth Factor Receptor. Target Oncol. 2024 May;19(3):333-342. doi: 10.1007/s11523-024-01051-2. Epub 2024 Mar 28. PMID 38546944